CLINICAL TRIAL: NCT06146803
Title: How Much the "Level of Resilience" Influences Self-care in a Group of Subjects Suffering From Heart Failure: Observational, Cross-sectional Study
Brief Title: the "Level of Resilience" Influencing Self-care in Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6079
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-11

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adaptation to the new health condition and self-care skills allow people to be able to adhere to the therapeutic treatment in the most correct way possible, but there are many cases in which subjects do not show adherence to it, and for this reason the risk increases to manifest acute complications and also to develop long-term ones

DETAILED DESCRIPTION:
Primary objective

-Evaluate levels of resilience in subjects suffering from heart failure.

Secondary objectives

* Evaluate the levels of self-care in subjects suffering from heart failure.
* Evaluate the correlation between the level of resilience and the level of self-care;
* Evaluate which characteristics positively influence the level of resilience and the degree of self-care of the person with heart failure.

Consecutive patients suffering from heart failure followed at the Cardiology department of the Agostino Gemelli IRCCS University Polyclinic Foundation of Rome will be included

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from heart failure;
* Subject aged between >18 years and <90 years;
* Ability to understand the Italian language;
* Clinical conditions that allow the questionnaire to be completed;
* Ability to provide written informed consent.

Exclusion Criteria:

* Subjects suffering from other forms of diabetes;
* Subjects suffering from serious psychiatric disorders;
* Serious clinical conditions that do not allow the questionnaire to be completed;
* Inability to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients suffering from heart failure followed at the Cardiology department of the Agostino Gemelli IRCCS University Polyclinic Foundation of Rome will be included
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate levels of resilience in subjects suffering from heart failure | 12 months

SECONDARY OUTCOMES:
Evaluate levels of self-care in subjects suffering from heart failure | 12 months
Evaluate the correlation between the level of resilience and the level of self-care | 12 months
Evaluate which characteristics positively influence the level of resilience and the degree of self-care of patients with heart failure | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCSS, Rome, RM, Italy